CLINICAL TRIAL: NCT05388994
Title: Effects of Exercise-related Irisin on Inflammation and Pain in Individuals With Osteoarthritis
Brief Title: Exercise-related Irisin on Inflammation and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Principal Investigator, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FiratUnive.
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Osteo Arthritis Knee; Pain; Inflammation
Keywords: Osteoarthritis; pain; irisin; inflammation; exercise
MeSH Terms: conditions — Pain; Inflammation; Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): The initial implementation for the 8-week combined exercise program consisted of a progressive aerobic exercise program with a lower extremity bike (Ergoline Ergoselect 200; Ergoline GMBH, Bitz, Germany). All sessions are individually supervised and conducted. Training intensity was started at 70% of maximum aerobic capacity and training intensity was increased by 5% of VO2peak every two weeks. Pedal speed was fixed at 50 rpm throughout 8 weeks of training. Exercise sessions; It started with a 5 minute warm-up period (30% of VO2peak), followed by a total of 40 minutes with a 30-minute load period and a 5-minute cool-down period (without resistance).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The initial implementation for the 8-week combined exercise program consisted of a progressive aerobic exercise program with a lower extremity bike (Ergoline Ergoselect 200; Ergoline GMBH, Bitz, Germany). All sessions are individually supervised and conducted. Training intensity was started at 70% of maximum aerobic capacity and training intensity was increased by 5% of VO2peak every two weeks. Pedal speed was fixed at 50 rpm throughout 8 weeks of training. Exercise sessions; It started with a 5 minute warm-up period (30% of VO2peak), followed by a total of 40 minutes with a 30-minute load period and a 5-minute cool-down period (without resistance).

SUMMARY:
Osteoarthritis (OA) is a chronic disease that usually starts with cartilage damage in weight-bearing joints and then causes pain and loss of function secondary to damage in surrounding tissues. Osteoarthritis, which is seen with a frequency of approximately 10% in men over the age of 60 and approximately 18% in women, ranks first among the diseases related to the joint. Many factors such as age, gender, obesity, physical activity, trauma, and genetic factors are involved in the etiology of the disease. In osteoarthritis, intra-articular production and destruction events can occur simultaneously, so it is a dynamic process. Among the joints in the lower and upper extremities, osteoarthritis is most common in the knee joint. Various approaches are used in the treatment, including drug therapy, hyaluronic acid injection, use of glucosamine and chondritis sulfate, exercises, physiotherapy applications, and diet applications for weight loss to reduce pain and increase physical function.

Physiotherapy and rehabilitation are important treatment options in OA. Generally, range of motion exercises, strengthening exercises, and endurance exercises are applied to patients. An exercise program can be as effective as an NSAID in reducing pain. Decreased quadriceps muscle strength is a finding seen in patients with symptomatic knee OA. In addition, aerobic exercise has the potential to improve cardiovascular fitness, many of the comorbidities often associated with OA, such as diabetes, hypertension, and obesity.

Because OA is a major public health problem, a less costly population-based approach is desirable. Therefore, the aim of this study was to investigate the effects of exercise-related irisin on inflammation and pain in patients with OA who underwent exercise.

DETAILED DESCRIPTION:
Osteoarthritis, which is seen with a frequency of approximately 10% in men over the age of 60 and approximately 18% in women, ranks first among the diseases related to the joint. Many factors such as age, gender, obesity, physical activity, trauma, and genetic factors are involved in the etiology of the disease. In osteoarthritis, intra-articular production and destruction events can occur simultaneously, so it is a dynamic process. Among the joints in the lower and upper extremities, osteoarthritis is most common in the knee joint. Various approaches are used in the treatment, including drug therapy, hyaluronic acid injection, use of glucosamine and chondritis sulfate, exercises, physiotherapy applications, and diet applications for weight loss to reduce pain and increase physical function.

The most important indicator of osteoarthritis is cartilage destruction. In general, the main factor that initiates cartilage damage is the abnormal mechanical forces that the joint is exposed to. It is thought that the most important factors in the pathogenesis of cartilage damage are chondrocytes, which are sensitive to mechanical loading. Chondrocytes additionally have the ability to produce and respond to inflammatory mediators. Chondrocytes secrete catabolic enzymes such as nitric oxide synthetase and cyclooxygenase, matrix metalloproteinases (MMP), disintegrin-metalloproteinase containing thrombospondin 1 domain (ADAMTS 4 and 5) and proinflammatory cytokines. is considered. In addition, prostaglandin E 2 (PGE 2) and nitric oxide (NO) have been described as effective mediators of inflammation and cartilage destruction. Proinflammatory cytokines [for example, interleukin-1 (IL-1), interleukin-6 (IL-6) and tumor necrosis factor-a (TNFα)] cyclooxygenase-2 (COX-2) and nitric oxide synthase (NOS), particularly NOS induces the expression of the inducible isoform (iNOS). COX-2 and iNOS are responsible for the increase in PGE 2 and NO levels, which play an important role in inflammation and pain. Therefore, it can be predicted that the severity of OA will be related to local prostanoid levels and/or other proinflammatory messengers.

Physiotherapy and rehabilitation is one of the important treatment options in OA. Generally, range of motion exercises, strengthening exercises and endurance exercises are applied to patients. An exercise program can be as effective as an NSAID in reducing pain. Decreased quadriceps muscle strength is a finding seen in patients with symptomatic knee OA. In addition, aerobic exercise has the potential to improve cardiovascular fitness, many of the comorbidities often associated with OA, such as diabetes, hypertension, and obesity.

In humans, increased levels of physical activity are generally associated with reduced concentrations of circulating proinflammatory mediators such as C-reactive protein and tumor necrosis factor a (TNFα). Interleukin-6 (IL-6), which is proinflammatory under certain conditions, is released at high levels from exercising muscles and has been shown to exert anti-inflammatory effects on TNFα and endotoxin-induced inflammation.

Irisin is an exercise-induced myokine that has attracted the attention of the scientific community for its potential thermogenic effect. It has been found that the release of irisin is stimulated by exercise in people who exercise for a certain period of time. However, studies on the effect of irisin on inflammatory and pain in individuals with OA have not been found in the literature. Because OA is a major public health problem, a less costly population-based approach is desirable. Therefore, the aim of this study was to investigate the effects of exercise-related irisin on inflammation and pain in patients with OA who underwent exercise.

In this study, patients who will be diagnosed with osteoarthritis by the Fırat University Training and Research Hospital, and orthopedic specialist will be evaluated prospectively. Patients; Before and after exercise, irisin value and C-Reactive Protein, Substance p, Interleukin-6, TNFalpha, Cyclooxygenase 2, Neuropeptide y, cartilage oligomeric matrix protein (COMP) and Matrix metalloproteinase 3 factors will be measured. In addition, as demographic characteristics of the patients; age, gender, body weight, height, occupation and education level of the patients, and the history of the disease will be taken. Orthopedic evaluation form; muscle strength, range of motion, gait analysis, pain status, contracture status, obesity status, the status of intracapsular structures, etc. information will be received.

With these data, it will be investigated whether the pain and inflammation values of the patients change with irisin before and after exercise, and which factors depend on it.

diagnosis of osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with osteoarthritis
* No knee joint contracture

Exclusion Criteria:

* Those with cardiopulmonary disease
* Individuals who exercise regularly
* Those who received intra-articular injection therapy in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-18 (Estimated); Primary Completion 2022-07-18 (Estimated); Study Completion 2022-08-18 (Estimated)

PRIMARY OUTCOMES:
Kellgren-Lawrence Scale | 8 weeks
  Radiologic examinations are the most important examination that gives us information in the diagnosis of gonarthrosis. AP and lateral radiographs taken by standing up give us precise information about the severity of the disease and the treatment to be planned. . In cases where the disease is more advanced, intra-knee joint mouse, subluxation and severe deformities can be seen. The Kellgren-Lawrence Scale, which was described in 1957, is used in radiological staging. Classification is made as 5 items. Stage 0: There is no sign of osteoarthritis.
  Stage 1: Suspected joint space narrowing and possible osteophyte formation. Stage 2: Definite osteophyte and possible joint space narrowing. Stage 3: Numerous osteophytes, definite narrowing of the joint space, sclerosis, and deformity of the bone boundaries may be present.
  Stage 4: Large osteophytes, severe narrowing of the joint space, severe sclerosis, and overt deformities of the bone margins.
Lequesne knee osteoarthritis severity index | 8 weeks
  he Lequesne knee osteoarthritis index (LDOI), which was defined in 1989, aims to measure the severity of osteoarthritis involvement in the knee joint. It questions pain and discomfort (5 questions), walking (2 questions), and activities in daily life (4 questions). The weight of the questions is different and the result is a score between 0 and 24.
WOMAC scale | 8 weeks
  The WOMAC scale is a measure of health status specific to osteoarthritis. It consists of three parts and 24 questions that assess clinically significant pain, stiffness, and physical function status in patients with knee or hip osteoarthritis. It can be completed in 5 minutes. Each question was scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated on its own and the total score ranges from 0 to 100. High scores indicate increased pain and stiffness, impaired physical function.
Irisin Hormone Analiz | 8 weeks
  Samples of venous blood were collected after overnight (12 h) fasting in the morning before and after the study from all patients. Venous blood was drawn using venipuncture and clotted for serum and centrifuged at 4000g for 5 minutes at 4°C. Serum samples then were aliquoted, and stored at -80°C until were assayed with enzyme-linked immunosorbent assay (ELISA) analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Furkan Bilek, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moffet H, Collet JP, Shapiro SH, Paradis G, Marquis F, Roy L. Effectiveness of intensive rehabilitation on functional ability and quality of life after first total knee arthroplasty: A single-blind randomized controlled trial. Arch Phys Med Rehabil. 2004 Apr;85(4):546-56. doi: 10.1016/j.apmr.2003.08.080. PMID 15083429
- [Background] Felson DT. An update on the pathogenesis and epidemiology of osteoarthritis. Radiol Clin North Am. 2004 Jan;42(1):1-9, v. doi: 10.1016/S0033-8389(03)00161-1. PMID 15049520
- [Background] Goldring MB, Marcu KB. Cartilage homeostasis in health and rheumatic diseases. Arthritis Res Ther. 2009;11(3):224. doi: 10.1186/ar2592. Epub 2009 May 19. PMID 19519926
- [Background] Goldring MB, Otero M, Plumb DA, Dragomir C, Favero M, El Hachem K, Hashimoto K, Roach HI, Olivotto E, Borzi RM, Marcu KB. Roles of inflammatory and anabolic cytokines in cartilage metabolism: signals and multiple effectors converge upon MMP-13 regulation in osteoarthritis. Eur Cell Mater. 2011 Feb 24;21:202-20. doi: 10.22203/ecm.v021a16. PMID 21351054
- [Background] Hedbom E, Hauselmann HJ. Molecular aspects of pathogenesis in osteoarthritis: the role of inflammation. Cell Mol Life Sci. 2002 Jan;59(1):45-53. doi: 10.1007/s00018-002-8404-z. PMID 11846032
- [Background] Raisz LG. Prostaglandins and bone: physiology and pathophysiology. Osteoarthritis Cartilage. 1999 Jul;7(4):419-21. doi: 10.1053/joca.1998.0230. PMID 10419786
- [Background] Abramson SB, Attur M, Amin AR, Clancy R. Nitric oxide and inflammatory mediators in the perpetuation of osteoarthritis. Curr Rheumatol Rep. 2001 Dec;3(6):535-41. doi: 10.1007/s11926-001-0069-3. PMID 11709117
- [Background] Jang D, Murrell GA. Nitric oxide in arthritis. Free Radic Biol Med. 1998 Jun;24(9):1511-9. doi: 10.1016/s0891-5849(97)00459-0. PMID 9641270
- [Background] Evans CH, Stefanovic-Racic M, Lancaster J. Nitric oxide and its role in orthopaedic disease. Clin Orthop Relat Res. 1995 Mar;(312):275-94. PMID 7543392
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] American College of Sports Medicine. Position Stand. Physical activity, physical fitness, and hypertension. Med Sci Sports Exerc. 1993 Oct;25(10):i-x. PMID 8231750
- [Background] Seals DR, Hagberg JM, Hurley BF, Ehsani AA, Holloszy JO. Effects of endurance training on glucose tolerance and plasma lipid levels in older men and women. JAMA. 1984 Aug 3;252(5):645-9. PMID 6376837
- [Background] You T, Nicklas BJ. Effects of exercise on adipokines and the metabolic syndrome. Curr Diab Rep. 2008 Feb;8(1):7-11. doi: 10.1007/s11892-008-0003-4. PMID 18366992
- [Background] Mathur N, Pedersen BK. Exercise as a mean to control low-grade systemic inflammation. Mediators Inflamm. 2008;2008:109502. doi: 10.1155/2008/109502. Epub 2009 Jan 11. PMID 19148295
- [Background] Palacios-Gonzalez B, Vadillo-Ortega F, Polo-Oteyza E, Sanchez T, Ancira-Moreno M, Romero-Hidalgo S, Meraz N, Antuna-Puente B. Irisin levels before and after physical activity among school-age children with different BMI: a direct relation with leptin. Obesity (Silver Spring). 2015 Apr;23(4):729-32. doi: 10.1002/oby.21029. PMID 25820255
- [Background] Duncan R, Peat G, Thomas E, Hay E, McCall I, Croft P. Symptoms and radiographic osteoarthritis: not as discordant as they are made out to be? Ann Rheum Dis. 2007 Jan;66(1):86-91. doi: 10.1136/ard.2006.052548. Epub 2006 Jul 28. PMID 16877532
- [Background] Lequesne MG, Mery C, Samson M, Gerard P. Indexes of severity for osteoarthritis of the hip and knee. Validation--value in comparison with other assessment tests. Scand J Rheumatol Suppl. 1987;65:85-9. doi: 10.3109/03009748709102182. PMID 3479839
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365